CLINICAL TRIAL: NCT02229604
Title: Electroacupuncture for Diminished Ovarian Reserve-a Cohort Study
Brief Title: Electroacupuncture for Diminished Ovarian Reserve
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guangan'men Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZ0708081
Record Dates: First submitted 2014-08-25; First posted 2014-09-01 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Irregular Menses
Keywords: electroacupuncture; diminished ovarian reserve; cohort study
MeSH Terms: conditions — Menstruation Disturbances | interventions — Acupuncture Therapy; Hormone Replacement Therapy; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EA group (Experimental): Patients choose this group will receive EA as a combination. Beside of EA, participants could receive oral medicine as the same as that of the drug group. The EA regimen has two point formulae, i.e. A (BL33) and B (ST25, EX-CA1 and RN4). The two formulae will be used alternatively. One session will last for 20 minutes, 5 sessions per week for the first 4 weeks and 3 sessions per week later (44 sessions in all).
  Interventions: Other: EA; Drug: HRT, DHEA and herb
- drug group (Active Comparator): Hormone replacement therapy (HRT), DHEA and herb decoction are allowed to be used for this group. Treatment course is not fixed. Immunosuppressive agents are not allowed.
  Interventions: Drug: HRT, DHEA and herb

INTERVENTIONS:
Other: EA — For BL33, insert the needle to the third posterior sacral foramina to a depth of 80-100mm. For ST25, EX-CA1 and RN4, the needle will be inserted vertically and quickly through the skin, and then slowly and vertically penetrate through the layer of fatty tissue, up into the muscles of the abdominal wall (until the moment of resistance is sensed on the tip of the needle and the participant feels a sting). The electric stimulator will be put on the BL33 and EX-CA1 with a continuous wave, 20 Hz, 1.0-4.0 mA.
  Other Names: acupuncture
  Arms: EA group
Drug: HRT, DHEA and herb — HRT, dehydroepiandrosterone (DHEA) and herb decoction could be used for this group. Time frame of treatment is not fixed. Herb decoction will be given to participants based on the principle of syndrome differentiation (a diagnosing method in Traditional Chinese Medicine).

SUMMARY:
Diminished ovarian reserve (DOR)is a disease can not be cured. Medicine for DOR includes dehydroepiandrosterone (DHEA), hormone replacement therapy (HRT), immunosuppressive agents and alternative therapy, etc. Electroacupuncture (EA) can help patients regain regular menses, increase the estradiol (E2) level and decrease the follicle-stimulating hormone (FSH) and decrease FSH/luteotropic (LH) ratio. In this cohort study, we aim to observe the effect of EA versus other therapies for DOR.

ELIGIBILITY:
Inclusion Criteria:

* Age younger than 40 yr
* 10IU/L ≤ FSH ≤ 40IU/L
* Volunteer to join the research and give the informed consent

Exclusion Criteria:

* A history of ovariectomy, receiving cytotoxic chemotherapy or irradiation
* Reproductive system infection or tumor
* Autoimmune disease
* Amenorrhea due to reproduction abnormality or pregnancy
* Patients can not adhere to treatment due to personal situation
* Patients have taken immunosuppressive agents in past 6 months
* receive treatment for less than 1 week before withdrawal

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change of FSH from baseline | baseline, week 12
  The follicle-stimulating hormone (FSH) will be tested at baseline and week 12

SECONDARY OUTCOMES:
change of FSH level from baseline | baseline, week 4, 8, 16, 20, and 24
  FSH will be tested at baseline and week 4, 8, 16, 20, and 24
changes in FSH/LH ratio, LH, and E2 from baseline | baseline, week 4, 8, 12, 16, 20, and 24
  FSH/LH ratio, LH, and E2 will be tested at baseline and week 4, 8, 12, 16, 20, and 24
change of symptom scale | baseline, week 12, week 24
  Symptoms need to be assessed include irritability and depression. A 4-point scale is used to evaluate the degree of symptoms (0 means "not at all" and 3 means "severe").
proportion of patients regaining regular menses | baseline, weeks 8, 12 and 24
  The proportion of patients regaining regular menses at week8, 12 and 24 will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Ph.D, Study Chair — Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Li Y, Chen R, Cui X, Yu J, Liu Z. Electroacupuncture for reproductive hormone levels in patients with diminished ovarian reserve: a prospective observational study. Acupunct Med. 2016 Oct;34(5):386-391. doi: 10.1136/acupmed-2015-011014. Epub 2016 May 13. PMID 27177929